CLINICAL TRIAL: NCT07207863
Title: The Cardiac and Panvascular Medicine Diagnosis and Treatment Center, People's Hospital of Xinjiang Uygur Autonomous Region,
Brief Title: Tianshan Community Cohort Establishment and Follow-up
Status: Recruiting | Type: Observational
Sponsor: People's Hospital of Xinjiang Uygur Autonomous Region (Other)
Collaborators: People's Hospital of Hotan Prefecture (Unknown); People's Hospital of Altay Prefecture (Unknown); Luopu County People's Hospital of Hotan Prefecture (Unknown); The First People's Hospital of Aksu Prefecture (Unknown); Karamay Central Hospital of Xinjiang (Unknown); People's Hospital of Kizilsu Kyrgyz Autonomous Prefecture (Unknown); The Second People's Hospital of Kashgar Prefecture (Unknown); RenJi Hospital (Other)
Responsible Party: Principal Investigator, Yining Yang, Prof., People's Hospital of Xinjiang Uygur Autonomous Region
Other Study IDs: Tianshan2025
Record Dates: First submitted 2025-09-27; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Cohort Study; Natural Population; Northwest Region of China

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During routine health checkups, 10 mL of EDTA-anticoagulated blood, 10 mL of urine, 10 g of feces and 2 mL of saliva are collected. Samples are transported to the Biobank of the People's Hospital of Xinjiang Uygur Autonomous Region for processing within 2 hours and subsequently stored at -80 °C in an ultra-low temperature freezer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This population-based cohort study on disease prevention and health promotion was established in northwest China, leveraging data from routine annual health examinations. Initiated in January 2016, the cohort enrolled nearly all residents aged 18 years and older who were registered at community healthcare centers. The program was developed to provide a comprehensive framework for disease prevention and community health promotion, with the aim of producing population-based evidence across a broad spectrum of diseases in the general population. At baseline, data were collected on participant demographics, medical and family histories, disability status, living environment, and blood biochemical parameters. Follow-up information is primarily obtained through chronic disease management programs, annual health examinations, and electrical health records. Cause-specific mortality is ascertained from local death registration systems. Biological specimens, questionnaire data, and electrical health records are systematically archived in the Biobank and Big Data Center of the People's Hospital of Xinjiang Uygur Autonomous Region.

DETAILED DESCRIPTION:
This research is conducted through population-based health examinations among residents in northwest China. By providing annual health assessments, structured health education, and community-based health promotion activities, the study aims to enhance health awareness, identify determinants of disease, implement targeted interventions to improve lifestyle behaviors, reduce modifiable risk factors, and promote overall community health.

The cohort integrates data from multiple sources- including health assessments, electronic health records, mortality registries, statistical yearbooks, and environmental datasets- encompassing a wide range of health-related information, such as demographics, lifestyle factors, family and personal medical histories, living conditions, enrollment in national public health services, physical examinations, laboratory tests, diagnostic assessments, disease outcomes, and cause-specific mortality. Event-driven follow-up data are obtained from 163 hospitals and 63 Traditional Chinese Medicine hospitals, covering all secondary and tertiary-level hospitals in the region. Inpatient data are systematically documented by qualified medical personnel and entered into an electronic health information system. All disease diagnoses are coded according to the 10th Revision of the International Classification of Diseases (ICD-10). Mortality data, including the timing and specific cause of death, are primarily obtained through local death registration systems.

ELIGIBILITY:
Inclusion Criteria:

1. Residents >=18y
2. Permanent residents or individuals who have lived in the region for more than 5 years and are enrolled in local social security medical insurance
3. Residents without severe physical disability and capable of normal communication
4. Residents whose diseases and deaths are monitored and managed by the local health authorities
5. Residents who voluntarily participate and provide written informed consent

Exclusion Criteria:

1. Temporary residents or floating population
2. Residents with severe health conditions that prevent participation in the study
3. Residents who are unwilling to undergo follow-up assessments for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible residents from routine annual health examinations.
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 20 years
  All-cause and cause-specific mortality during follow-up
Cardiovascular diseases | 20 years
  Incident disease during follow-up
Digestive diseases | 20 years
  Incident disease during follow-up
Endocrine diseases | 20 years
  Incident disease during follow-up
Infections diseases | 20 years
  Incident disease during follow-up
Benign neoplasm or Carcinoma in situ | 20 years
  Incident disease during follow-up
Cancers | 20 years
  Incident disease during follow-up
Genitourinary diseases | 20 years
  Incident disease during follow-up
Haematological or immunological diseases | 20 years
  Incident disease during follow-up
Musculoskeletal diseases | 20 years
  Incident disease during follow-up
Neurological diseases | 20 years
  Incident disease during follow-up
Psychiatric diseases | 20 years
  Incident disease during follow-up
Respiratory diseases | 20 years
  Incident disease during follow-up
Ocular diseases | 20 years
  Incident disease during follow-up
Dermatological diseases | 20 years
  Incident disease during follow-up
Ear and mastoid disorders | 20 years
  Incident disease during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Yining Yang, Prof., Principal Investigator — People's Hospital of Xinjiang Uygur Autonomous Region
Locations (1):
- People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: No